CLINICAL TRIAL: NCT03485911
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Two Dose Levels of BCX7353 as an Oral Treatment for the Prevention of Attacks in Subjects With Hereditary Angioedema
Brief Title: Efficacy and Safety Study of BCX7353 as an Oral Treatment for the Prevention of Attacks in HAE
Acronym: APeX-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BCX7353-302
Record Dates: First submitted 2018-03-15; First posted 2018-04-03 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-05

CONDITIONS: Hereditary Angioedema; HAE
Keywords: BCX7353; Berotralstat
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only Part 1 and Part 2 were blinded. As part 3 was open-label, no blinding was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BCX7353 110 mg once daily (Experimental): BCX7353 administered as oral capsules once daily
  Interventions: Drug: BCX7353 capsules
- BCX7353 150 mg once daily (Experimental): BCX7353 administered as oral capsules once daily
  Interventions: Drug: BCX7353 capsules
- Placebo (Placebo Comparator): Matching placebo administered as oral capsules once daily
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: BCX7353 capsules — BCX7353 oral capsules administered once daily
  Other Names: Berotralstat
  Arms: BCX7353 110 mg once daily; BCX7353 150 mg once daily
Drug: Placebo oral capsule — Matching oral capsules administered once daily
  Arms: Placebo

SUMMARY:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of oral BCX7353 in preventing acute angioedema attacks in patients with Type I and Type II HAE.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of hereditary angioedema Type 1 or Type 2, defined as having a C1-INH functional level and a C4 level below the lower limit of the normal (LLN) reference range, as assessed during the Screening period.
* Subject weight of ≥ 40 kg
* Access to and ability to use one or more acute medications approved by the relevant competent authority for the treatment of acute attacks of HAE
* Subjects must be medically appropriate for on-demand treatment as the sole medicinal management for their HAE during the study.
* Subjects must have a specified number of investigator-confirmed attacks during the run-in period of a maximum of 56 days from the Screening visit.
* Acceptable effective contraception
* Written informed consent

Key Exclusion Criteria:

* Pregnancy or breast-feeding
* Any clinically significant medical condition or medical history that, in the opinion of the Investigator or Sponsor, would interfere with the subject's safety or ability to participate in the study
* Any laboratory parameter abnormality that, in the opinion of the Investigator, is clinically significant and relevant for this study
* Severe hypersensitivity to multiple medicinal products or severe hypersensitivity/ anaphylaxis with unclear etiology
* Use of C1-INH within 14 days or use of androgens or tranexamic acid within 28 days prior to the Screening visit for prophylaxis of HAE attacks, or initiation of these drugs during the study
* Current participation in any other investigational drug study or received another investigational drug within 30 days of the Screening visit
* Prior enrollment in a BCX7353 study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 121 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Zuraw, MD, Principal Investigator — UC San Diego School of Medicine, US HAE Angioedema Center
Locations (47):
- United States (27):
  - Study center, Birmingham, Alabama
  - Study center, Scottsdale, Arizona
  - Study center, Little Rock, Arkansas
  - Study Center, San Diego, California
  - Study center, Santa Monica, California
  - Study Center, Walnut Creek, California
  - Study center, Colorado Springs, Colorado
  - Study Center, Tampa, Florida
  - Study center, Chevy Chase, Maryland
  - Study Center, Boston, Massachusetts
  - Study Center, Ann Arbor, Michigan
  - Study center, Plymouth, Minnesota
  - Study Center, St Louis, Missouri
  - Study center, Belleville, New Jersey
  - Study Center, Fair Lawn, New Jersey
  - Study center, Piscataway, New Jersey
  - Study Center, New York, New York
  - Study Site, Charlotte, North Carolina
  - Study Center, Durham, North Carolina
  - Study Center, Cincinnati, Ohio
  - Study center, Columbus, Ohio
  - Study center, Clackamas, Oregon
  - Study Center, Hershey, Pennsylvania
  - Study center, Austin, Texas
  - Study center, Dallas, Texas
  - Study Center, San Antonio, Texas
  - Study Center, Spokane, Washington
- Study Center, Vienna, Austria
- Canada (3):
  - Study Center, Ottawa, Ontario
  - Study Center, Toronto, Ontario
  - Study Center, Québec
- Czechia (2):
  - Study Center, Brno
  - Study Center, Pilsen
- France (2):
  - Study Center, Grenoble
  - Study Center, Paris
- Germany (2):
  - Study Center, Berlin
  - Study Center, Frankfurt
- Study Center, Budapest, Hungary
- Study Center, Skopje, North Macedonia
- Study Center, Sângeorgiu de Mureș, Jud. Mureș, Romania
- Spain (3):
  - Study Center, Barcelona
  - Study Center, Madrid
  - Study Center, Seville
- United Kingdom (4):
  - Study Center, Cambridge
  - Study Center, Frimley
  - Study Center, London
  - Study Center, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farkas H, Balla Z. A review of berotralstat for the treatment of hereditary angioedema. Expert Rev Clin Immunol. 2023 Feb;19(2):145-153. doi: 10.1080/1744666X.2023.2150611. Epub 2022 Nov 29. PMID 36408587
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Wedner HJ, Aygoren-Pursun E, Bernstein J, Craig T, Gower R, Jacobs JS, Johnston DT, Lumry WR, Zuraw BL, Best JM, Iocca HA, Murray SC, Desai B, Nagy E, Sheridan WP, Kiani-Alikhan S. Randomized Trial of the Efficacy and Safety of Berotralstat (BCX7353) as an Oral Prophylactic Therapy for Hereditary Angioedema: Results of APeX-2 Through 48 Weeks (Part 2). J Allergy Clin Immunol Pract. 2021 Jun;9(6):2305-2314.e4. doi: 10.1016/j.jaip.2021.03.057. Epub 2021 Apr 15. PMID 33866032
- [Derived] Zuraw B, Lumry WR, Johnston DT, Aygoren-Pursun E, Banerji A, Bernstein JA, Christiansen SC, Jacobs JS, Sitz KV, Gower RG, Gagnon R, Wedner HJ, Kinaciyan T, Hakl R, Hanzlikova J, Anderson JT, McNeil DL, Fritz SB, Yang WH, Tachdjian R, Busse PJ, Craig TJ, Li HH, Farkas H, Best JM, Clemons D, Cornpropst M, Dobo SM, Iocca HA, Kargl D, Nagy E, Murray SC, Collis P, Sheridan WP, Maurer M, Riedl MA. Oral once-daily berotralstat for the prevention of hereditary angioedema attacks: A randomized, double-blind, placebo-controlled phase 3 trial. J Allergy Clin Immunol. 2021 Jul;148(1):164-172.e9. doi: 10.1016/j.jaci.2020.10.015. Epub 2020 Oct 21. PMID 33098856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with HAE Type 1 or Type 2 were eligible for the study following assessment of data obtained from screening procedures, including demonstration of a minimum number of qualifying HAE attacks documented during a prospective run-in period of 14 to 56 days from the date of the screening visit. Randomization was stratified by the HAE attack rate over the period between screening and randomization (≥ 2 attacks per month vs. < 2 attacks per month).
Groups:
- Treatment Group 1 (110 mg Berotralstat QD): Parts 1 and 2: two 55 mg capsules of berotralstat QD × 48 weeks. Part 3: 150 mg berotralstat QD.
- Treatment Group 2 (150 mg Berotralstat QD): Parts 1 and 2: two 75 mg capsules of berotralstat QD × 48 weeks. Part 3: 150 mg berotralstat QD.
- Treatment Group 3a: Subjects were treated with placebo in Part 1 and 110 mg berotralstat in part 2. In part 3 subjects were treated with 150 mg berotralstat QD.
- Treatment Group 3b: Subjects were treated with placebo in Part 1 and 150 mg berotralstat QD in part 2 and 3.
Period: Part 1
Arm/Group | Treatment Group 1 (110 mg Berotralstat QD) | Treatment Group 2 (150 mg Berotralstat QD) | Treatment Group 3a | Treatment Group 3b
Started | 41 | 40 | 20 | 20
Completed | 37 | 37 | 17 | 17
Not Completed | 4 | 3 | 3 | 3
Not completed — Perceived lack of efficacy | 1 | 1 | 2 | 0
Not completed — Subject withdrew consent | 0 | 1 | 0 | 1
Not completed — Lab abnormalities/AEs | 3 | 1 | 1 | 0
Not completed — Withdrew Consent prior to dosing | 0 | 0 | 0 | 1
Not completed — Other NOS | 0 | 0 | 0 | 1
Period: Part 2
Arm/Group | Treatment Group 1 (110 mg Berotralstat QD) | Treatment Group 2 (150 mg Berotralstat QD) | Treatment Group 3a | Treatment Group 3b
Started | 37 | 37 | 17 | 17
Completed | 28 | 31 | 15 | 14
Not Completed | 9 | 6 | 2 | 3
Not completed — Perceived lack of efficacy | 5 | 3 | 0 | 2
Not completed — Subject withdrew consent | 1 | 0 | 2 | 1
Not completed — Lab abnormalities/AEs | 1 | 2 | 0 | 0
Not completed — Other NOS | 0 | 1 | 0 | 0
Not completed — Intercurrent illness/new medical condition | 1 | 0 | 0 | 0
Not completed — Investigator judgement | 1 | 0 | 0 | 0
Period: Part 3
Arm/Group | Treatment Group 1 (110 mg Berotralstat QD) | Treatment Group 2 (150 mg Berotralstat QD) | Treatment Group 3a | Treatment Group 3b
Started | 26 (Two subjects completed Part 2, but did not continue treatment in Part 3 due to: * Subject non-compliance with study drug (1 subject) * Other (1 subject)) | 26 (Five subjects completed Part 2, but did not continue treatment in Part 3 due to: * Perceived lack of efficacy (2 subjects) * Subject withdrew consent (1 subject) * Other (2 subjects)) | 15 | 14
Completed | 7 | 4 | 5 | 4
Not Completed | 19 | 22 | 10 | 10
Not completed — Perceived lack of efficacy | 2 | 2 | 2 | 0
Not completed — Subject withdrew consent | 1 | 4 | 0 | 1
Not completed — Lab abnormalities/AEs | 1 | 1 | 0 | 2
Not completed — Other NOS | 1 | 1 | 0 | 0
Not completed — Intercurrent illness/new medical condition | 0 | 1 | 1 | 0
Not completed — Sponsor discontinuation | 1 | 0 | 0 | 0
Not completed — Berotralstat provided by alternative means | 13 | 13 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Part 1: Berotralstat 110 mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD for 24 weeks.
- Part 1: Berotralstat 150 mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD for 24 weeks.
- Part 1: Placebo: Placebo administered as two 2 matching capsules, orally QD for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Berotralstat 110 mg Once Daily | Part 1: Berotralstat 150 mg Once Daily | Part 1: Placebo | Total
Number analyzed (Participants) | 41 | 40 | 40 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (17.51) | 40.0 (13.98) | 44.5 (14.12) | 41.6 (15.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 27 | 80
  Male | 11 | 17 | 13 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 39 | 38 | 38 | 115
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 38 | 38 | 37 | 113
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 3 | 3 | 10
  Austria | 1 | 2 | 1 | 4
  Romania | 0 | 1 | 0 | 1
  Hungary | 2 | 0 | 0 | 2
  United States | 28 | 24 | 25 | 77
  Czechia | 2 | 3 | 3 | 8
  North Macedonia | 0 | 1 | 1 | 2
  United Kingdom | 1 | 4 | 2 | 7
  France | 2 | 0 | 1 | 3
  Germany | 1 | 2 | 2 | 5
  Spain | 0 | 0 | 2 | 2
Baseline Investigator-confirmed attack rate [Count of Participants; unit: Participants] — Population: Safety Population. One subject from ITT population, randomised to the placebo group, was not dosed
  Participants
    ≥ 2 HAE attacks/month: number analyzed (Participants) | 41 | 40 | 39 | 120
    ≥ 2 HAE attacks/month | 28 | 30 | 27 | 85
    < 2 HAE attacks/month: number analyzed (Participants) | 41 | 40 | 39 | 120
    < 2 HAE attacks/month | 13 | 10 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Part 1: The Rate of Investigator-confirmed HAE Attacks During Dosing in the Entire 24-week Treatment Period (Day 1 to Day 168)
Description: Treatment comparisons between each berotralstat dose and placebo in the rate of investigator-confirmed HAE attacks during the Part 1 dosing period were analyzed using a negative binomial model. The number of investigator-confirmed attacks was included as the dependent variable, the treatment was included as a fixed effect, the stratification variable (baseline attack rate) was included as a covariate, and the logarithm of duration on treatment was included as an offset variable. The estimated attack rate for each treatment group, the treatment differences expressed as the attack rate ratio (berotralstat over placebo rate ratio), and the associated 95% confidence intervals (CIs) were provided from the negative binomial model.
Time Frame: 24 weeks
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy and health outcomes data.
Measure: Number; unit: HAE attack rate per 28 days
Groups:
- Berotralstat 110 mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD for 24 weeks.
- Berotralstat 150 mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD for 24 weeks.
- Placebo: Placebo administered as two matching capsules, orally QD for 24 weeks.
Arm/Group | Berotralstat 110 mg Once Daily | Berotralstat 150 mg Once Daily | Placebo
Number analyzed (Participants) | 41 | 40 | 40
HAE attack rate per 28 days | 1.65 | 1.31 | 2.35
Statistical Analysis 1: Comparison: Berotralstat 110 mg Once Daily vs Placebo; Test type: Superiority; p = 0.024, negative binomial regression model; negative binomial regression model = 30.0, 95% CI 2-sided [4.6 to 48.7]
Statistical Analysis 2: Comparison: Berotralstat 150 mg Once Daily vs Placebo; Test type: Superiority; p < 0.001, negative binomial regression model; negative binomial regression model = 44.2, 95% CI 2-sided [23.0 to 59.5]

2. Primary Outcome: Part 2 & 3: To Evaluate the Long-term Safety and Tolerability of Berotralstat 110 and 150 mg in Subjects With HAE
Description: The safety data was assessed for the safety population, for subjects who entered Part 2 and Part 3, and includes TEAEs that began in Part 2 or 3, respectively, for these subjects. Safety data for Part 2 and Part 3 is combined to clearly show TEAEs occurring in subjects as the proceeded through the 2 study parts. TEAEs are defined as AEs that occurred on or after first dose of study treatment, whether in Part 1 or 2, and were assigned to the relevant treatment depending on when the TEAE began (Part 2 or Part 3 treatment). No statistical analysis was performed on this safety data.
Time Frame: Part 2: 24 weeks (Days 169 to 337). Part 3: 48 weeks (Days 338 to 674).
Population: The safety population included all subjects who received at least 1 capsule of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: 110mg Berotralstat: Subjects were treated with 110 mg berotralstat QD in part 2
- Part 2: 110mg Berotralstat After Placebo: Subjects were treated with 110 mg berotralstat QD in part 2, following prior treatment with placebo in part 1.
- Part 2: 150mg Berotralstat: Subjects were treated with 150 mg berotralstat QD in part 2
- Part 2: 150mg Berotralstat Following Placebo: Subjects were treated with 150 mg berotralstat QD in part 2, following prior treatment with placebo in part 1.
- Part 3: Berotralstat: Subjects were treated with 150 mg berostralstat QD in part 3.
Arm/Group | Part 2: 110mg Berotralstat | Part 2: 110mg Berotralstat After Placebo | Part 2: 150mg Berotralstat | Part 2: 150mg Berotralstat Following Placebo | Part 3: Berotralstat
Number analyzed (Participants) | 37 | 17 | 37 | 17 | 81
Participants
  TEAE | 22 | 13 | 27 | 12 | 67
  Drug-related TEAE | 4 | 5 | 7 | 7 | 12
  TESAE | 0 | 0 | 1 | 1 | 7
  Drug-related TESAE | 0 | 0 | 0 | 0 | 0
  DMID grade 3 or 4 TEAE | 1 | 1 | 2 | 1 | 10
  Drug-related DMID grade 3 or 4 TEAE | 0 | 0 | 1 | 0 | 1
  TEAE leading to interruption of study drug | 0 | 1 | 2 | 1 | 5
  TEAE leading to discontinuation of study drug | 1 | 0 | 2 | 2 | 3
  Drug-related investigator-identified rash | 0 | 0 | 1 | 0 | 0
  GI abdominal-related TEAE | 5 | 4 | 10 | 9 | 18
  GI abdominal-related TEAE -study drug discontinued | 1 | 0 | 1 | 1 | 2

3. Secondary Outcome: Part 1: Change From Baseline in Angioedema Quality of Life Questionnaire at Week 24 (Total Score)
Description: Change in Quality of Life, on a 1-100 scale, where higher scores indicate more impairment and a decrease (change with a negative value) in AE-QoL questionnaire scores indicates an improvement in the subject's QoL. The minimum clinically important difference (MCID) for the AE-QoL questionnaire is -6 (total score). The AE-QoL is only validated for adults; however, data were collected on all adult and adolescent study subjects.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: AE-QoL Total Score Change from baseline
Arm/Group | Berotralstat 110 mg Once Daily | Berotralstat 150 mg Once Daily | Placebo
Number analyzed (Participants) | 40 | 38 | 36
AE-QoL Total Score Change from baseline | -12.46 (2.530) | -14.59 (2.592) | -9.69 (2.643)
Statistical Analysis 1: Comparison: Berotralstat 110 mg Once Daily vs Placebo; Numerical difference in change from baseline of AE-QoL total score between treatment groups; Test type: Superiority; p = 0.453, mixed-model repeated measures analysis; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-10.08 to 4.53]
Statistical Analysis 2: Comparison: Berotralstat 150 mg Once Daily vs Placebo; Numerical difference in change from baseline of AE-QoL total score between treatment groups; Test type: Superiority; p = 0.188, mixed-model repeated measures analysis; Mean Difference (Final Values) = -4.90, 95% CI 2-sided [-12.23 to 2.43]

4. Secondary Outcome: Part 1: Proportion of Days With Angioedema Symptoms Through 24 Weeks
Description: Assessment of proportion of days subjects had angioedema symptoms from expert-confirmed HAE attacks during Part 1.
Time Frame: 24 weeks
Population: The ITT population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy and health outcomes data. Data were analyzed according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Proportion days with angioedema symptoms
Arm/Group | Berotralstat 110 mg Once Daily | Berotralstat 150 mg Once Daily | Placebo
Number analyzed (Participants) | 41 | 40 | 40
Proportion days with angioedema symptoms | 0.134 (0.0191) | 0.119 (0.0194) | 0.197 (0.0196)
Statistical Analysis 1: Comparison: Berotralstat 110 mg Once Daily vs Placebo; Numerical differences from the placebo treatment in the LSM proportion of the 169 days of treatment with angioedema symptoms. In the event that the first secondary endpoint did not meet statistical significance in the hierarchical testing scheme, testing of the second secondary endpoint of proportion of days with angioedema symptoms through 24 weeks for statistical significance would not be completed. P-values that are reported are nominal; Test type: Superiority; p = 0.025, ANCOVA; Difference in Least Square Means = -0.062, 95% CI 2-sided [-0.117 to -0.008]
Statistical Analysis 2: Comparison: Berotralstat 150 mg Once Daily vs Placebo; Numerical differences from the placebo treatment in the LSM proportion of the 169 days of treatment with angioedema symptoms. In the event that the first secondary endpoint did not meet statistical significance in the hierarchical testing scheme, testing of the second secondary endpoint of number and proportion of days with angioedema symptoms through 24 weeks for statistical significance would not be completed. P-values that are reported are nominal; Test type: Superiority; p = 0.006, ANCOVA; Difference in Least Square Means = -0.078, 95% CI 2-sided [-0.133 to -0.023]

5. Secondary Outcome: Part 1: Rate of Expert-confirmed Angioedema Events During Dosing in the Effective Treatment Period
Description: The rate of expert-confirmed HAE attacks for the effective treatment period gives an analysis of the efficacy of active treatment after berotralstat had reached steady-state concentrations, given the effective half-life of 150 mg berotralstat in Study BCX7353-106 (Study 106) of 89 hours.
Time Frame: Day 8 through to 24 weeks (or or the last dose date/time in Part 1 + 24 hours for subjects who discontinued drug in Part 1)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: HAE attack rate per 28 days
Arm/Group | Berotralstat 110 mg Once Daily | Berotralstat 150 mg Once Daily | Placebo
Number analyzed (Participants) | 41 | 40 | 40
HAE attack rate per 28 days | 1.918 (1.7345) | 1.552 (1.6390) | 2.490 (1.6135)
Statistical Analysis 1: Comparison: Berotralstat 110 mg Once Daily vs Placebo; In the event that the first secondary endpoint did not meet statistical significance in the hierarchical testing scheme, testing of the third secondary endpoint of rate of expert-confirmed HAE attacks during dosing in the effective treatment period for statistical significance would not be completed. P-values reported are nominal; Test type: Superiority; p = 0.026, negative binomial regression model; negative binomial regression model = 30.4, 95% CI 2-sided [4.3 to 49.3]
Statistical Analysis 2: Comparison: Berotralstat 150 mg Once Daily vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.001, negative binomial regression model; negative binomial regression model = 46.5, 95% CI 2-sided [25.6 to 61.5]

6. Secondary Outcome: Part 2: To Assess the Effectiveness of Berotralstat Over a 24- to 48 Week Period
Description: Monthly Attack Rate was defined as the total number of investigator-confirmed HAE attacks experienced during the treatment period adjusted for the length of a month (defined as 28 days) and the number of days the subject was on treatment during that month. The end of Month 6 was defined as the start of Part 2 treatment.
  Baseline investigator-confirmed attack rate was defined as the total number of investigator-confirmed HAE attacks experienced in the period between screening and first dose of study drug adjusted for the length of a month (defined as 28 days) and the number of days during that period.
Time Frame: 24 weeks (Days 169 to 337)
Population: The intent to treat (ITT) population included all randomized subjects, regardless of whether study treatment was administered. This population was the primary population for the analysis of the efficacy data. The numbers analysed reflect participants providing details of HAE attacks via the study diary each month during part 2.
Measure: Mean (Standard Deviation); unit: HAE attack rate-change from baseline
Arm/Group | Part 2: 110mg Berotralstat | Part 2: 150mg Berotralstat
Number analyzed (Participants) | 53 | 51
HAE attack rate-change from baseline
  Month 6 | -1.383 (1.7289) | -1.593 (1.6581)
  Month 7: number analyzed (Participants) | 39 | 38
  Month 7 | -1.229 (1.8158) | -1.903 (1.7402)
  Month 12: number analyzed (Participants) | 32 | 32
  Month 12 | -1.543 (1.6539) | -1.910 (1.5330)

7. Secondary Outcome: To Evaluate Angioedema Quality of Life Questionnaire (Total Score) Following Berotralstat Administration for up to 144 Weeks
Description: Angioedema-specific QoL was assessed by the AE-QoL, consisting of 4 domains (i.e., functioning, fatigue/mood, fears/shame, and nutrition) and a total score. The AE-QoL scores range from 0 points (best QoL) to 100 points (worst QoL). A decrease (change with a negative value) in AE-QoL questionnaire scores indicates an improvement in the subject's QoL. The minimum clinically important difference (MCID) for the AE-QoL questionnaire is -6 (total score). The AE-QoL was completed by the subjects at each visit starting at baseline, and questions were answered with regard to the previous 28 days. For subjects who received active treatment following placebo, visits were adjusted according to the date of the first dose of active treatment.
Time Frame: Up to 144 weeks
Population: The ITT population included all randomized subjects, regardless of study treatment administration. Subjects in the 2 berotralstat treatment arms included those previously treated with placebo in part 1; for these subjects, visits were adjusted according to the date of 1st dose of active treatment. The variation in number of subjects analysed at each study visit reflects subject withdrawal prior to study completion and the number of subjects completing the AE-QoL questionnaire.
Measure: Mean (Standard Deviation); unit: AE-QoL score - change from baseline
Groups:
- Berotralstat 110/150 mg Once Daily: Berotralstat administered as two 55mg capsules, orally QD, until transitioned to 150 mg QD dose in Part 3.
- Berotralstat 150 mg Once Daily: Berotralstat administered as two 75mg capsules, orally QD
- Placebo: Placebo administered as two matching capsules, orally QD for 24 weeks in Part 1.
Arm/Group | Berotralstat 110/150 mg Once Daily | Berotralstat 150 mg Once Daily | Placebo
Number analyzed (Participants) | 58 | 55 | 39
AE-QoL score - change from baseline
  Week 4 | -5.85 (15.478) | -9.70 (15.346) | -7.762 (15.098)
  Week 8 | -10.58 (15.968) | -13.09 (19.064) | -11.33 (16.732)
  Week 12: number analyzed (Participants) | 57 | 53 | 38
  Week 12 | -11.51 (14.354) | -13.95 (17.652) | -10.63 (18.376)
  Week 18: number analyzed (Participants) | 41 | 38 | 36
  Week 18 | -9.97 (16.809) | -15.13 (14.946) | -12.48 (19.752)
  Week 24: number analyzed (Participants) | 56 | 53 | 36
  Week 24 | -9.80 (16.145) | -12.81 (19.181) | -12.51 (20.371)
  Week 48: number analyzed (Participants) | 48 | 47 | 0
  Week 48 | -10.19 (14.128) | -13.78 (16.219) |
  Week 72: number analyzed (Participants) | 39 | 34 | 0
  Week 72 | -12.34 (16.909) | -13.02 (16.276) |
  Week 96: number analyzed (Participants) | 37 | 31 | 0
  Week 96 | -12.81 (16.593) | -17.92 (17.161) |
  Week 120: number analyzed (Participants) | 32 | 26 | 0
  Week 120 | -15.24 (18.026) | -17.24 (14.943) |
  Week 144: number analyzed (Participants) | 16 | 14 | 0
  Week 144 | -11.29 (17.165) | -11.65 (16.558) |

8. Secondary Outcome: To Evaluate Treatment Satisfaction Questionnaire for Medication (TSQM) Following Berotralstat Administration for up to 144 Weeks
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) was completed by subjects at baseline and at each study visit until the end of the study. TSQM scores consisted of 14 items of which 13 items were made up of 3 specific scales (Effectiveness, Side Effects, and Convenience) and 1 global satisfaction scale (Global Satisfaction). At baseline, TSQM questionnaires were completed based on subject's satisfaction with usual medications. At all other time points for collection of TSQM, subjects were asked about their level of satisfaction or dissatisfaction with the study drug. Scales scores were calculated for each scale and were transformed into scores ranging from 0 to 100, with higher scores indicating higher satisfaction. TSQM score and corresponding change from baseline values were calculated at each visit. For subjects who received active treatment following placebo, visits were adjusted according to the date of the first dose of active treatment.
Time Frame: Up to 144 weeks
Population: The ITT population included all randomized subjects, regardless of study treatment administration. Subjects in the 2 berotralstat treatment arms included those previously treated with placebo in part 1; for these subjects, visits were adjusted according to the date of 1st dose of active treatment. The variation in number of subjects analysed at each study visit reflects subject withdrawal prior to study completion and the number of subjects completing the TSQM questionnaire.
Measure: Mean (Standard Deviation); unit: TSQM Global score - change from baseline
Arm/Group | Berotralstat 110/150 mg Once Daily | Berotralstat 150 mg Once Daily | Placebo
Number analyzed (Participants) | 57 | 54 | 39
TSQM Global score - change from baseline
  Week 4 | -1.3 (31.75) | 2.4 (31.91) | -18.1 (35.44)
  Week 8: number analyzed (Participants) | 57 | 54 | 38
  Week 8 | 4.3 (31.51) | 2.1 (31.66) | -19.2 (40.41)
  Week 12: number analyzed (Participants) | 57 | 52 | 38
  Week 12 | 4.4 (33.03) | 4.3 (31.32) | -21.1 (44.15)
  Week 18: number analyzed (Participants) | 40 | 36 | 34
  Week 18 | -1.8 (33.02) | -3.8 (32.69) | -18.9 (39.59)
  Week 24: number analyzed (Participants) | 56 | 52 | 35
  Week 24 | 3.1 (33.69) | 2.9 (33.96) | -20.8 (42.52)
  Week 48: number analyzed (Participants) | 48 | 45 | 0
  Week 48 | 5.4 (31.52) | 6.7 (28.87) |
  Week 72: number analyzed (Participants) | 39 | 32 | 0
  Week 72 | 11.0 (30.43) | 10.9 (22.88) |
  Week 96: number analyzed (Participants) | 37 | 30 | 0
  Week 96 | 13.9 (30.16) | 14.5 (22.31) |
  Week 120: number analyzed (Participants) | 31 | 26 | 0
  Week 120 | 12.7 (29.55) | 14.6 (20.75) |
  Week 144: number analyzed (Participants) | 16 | 14 | 0
  Week 144 | 4.5 (39.11) | 8.7 (22.79) |

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were assessed and recorded from the time that the Informed consent form was signed through the last follow-up visit, approximately 3 weeks following the last dose of study drug, or until the AE was resolved or the subject was in a clinically stable condition with regards to the AE.
Description: AE data is presented for patients from the Safety Population; i.e. those who received at least one dose of study drug. AEs were assigned to the relevant treatment (i.e., 110 mg berotralstat, 150 mg berotralstat, placebo) depending on when the AE began relative study drug administration.
Groups:
- Berotralstat 110mg Once Daily: Berotralstat administered as either two 55mg capsules, orally QD
- Berotralstat 150mg Once Daily: Berotralstat administered as either two 75mg capsules, orally QD
- Placebo: Placebo administered as two 2 matching capsules, orally QD
Arm/Group | Berotralstat 110mg Once Daily | Berotralstat 150mg Once Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/58 | 0/39
Serious Adverse Events (participants affected / at risk) | 5/57 | 5/58 | 2/39
Other Adverse Events (participants affected / at risk) | 56/58 | 53/57 | 30/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berotralstat 110mg Once Daily (N=57) | Berotralstat 150mg Once Daily (N=58) | Placebo (N=39)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Medical observation (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Berotralstat 110mg Once Daily (N=58) | Berotralstat 150mg Once Daily (N=57) | Placebo (N=39)
Nausea (Gastrointestinal disorders) | 10 (12) | 11 (16) | 7 (8)
Vomiting (Gastrointestinal disorders) | 5 (7) | 9 (14) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 7 (9) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 8 (12) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (8) | 10 (15) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (7) | 8 (10) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 6 (6) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 4 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (33) | 19 (46) | 9 (15)
Upper respiratory tract infection (Infections and infestations) | 8 (13) | 9 (10) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 2 (2)
Fatigue (General disorders) | 4 (4) | 5 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (3) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (3) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 4 (8) | 3 (3) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 7 (12) | 2 (5) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 4 (5) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03485911/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT03485911/SAP_001.pdf